CLINICAL TRIAL: NCT03690505
Title: Assessment of the Knowledge and Needs of Patients With AMD Before a Therapeutic Patient Education Program is Put in Place
Acronym: DEMELE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I16027/DEMELE
Record Dates: First submitted 2018-09-13; First posted 2018-10-01 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment (Other): Assessment of the Knowledge and Needs of Patients With AMD Before a Therapeutic Patient Education Program is Put in Place
  Interventions: Behavioral: Interviews

INTERVENTIONS:
Behavioral: Interviews — informant-based questionnaire semi-structured individual interviews focus group interviews

SUMMARY:
Age-related macular degeneration (AMD) is a disease that blurs the sharp, central vision you need for "straight-ahead" activities such as reading, sewing, and driving. AMD affects the macula, the part of the eye that allows you to see fine detail

The purpose of the study is to describe in patients with AMD and depending on the nature of their pathology (neovascular or atrophic):

(i) knowledge about their pathology (risk factors, symptoms, treatments, self-monitoring tool), (ii) their needs and (iii) impact on their daily lives

This study is to make an inventory of the knowledge of patients with AMD about their disease and risk factors using a questionnaire (Appendix 1) and to identify their needs, the impact of the disease on their daily lives during individual interviews by raising the recurrent data and confronting them during the focus group. The information gathered will enable the construction of a therapeutic education program for better patient care and to strengthen the patient's capacities so that he becomes an actor in his change throughout his care project.

This a 3 steps study:

1. 200 patients will be enrolled and answer a questionnaire on knowledge of the disease
2. Two groups of 20 patients will be selected to participate to a semi-structured individual interviews
3. Two focus groups of 10 patients will be organized to assess needs, expectations, satisfactions or to better understand opinions, motivations or behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Patient with AMD (neovascular and atrophic) whatever the stage of the disease
* Patient over 50
* Patient affiliated to a social security scheme
* Written informed consent of the patient

Exclusion Criteria:

* Patient unable to understand the information, fill out the questionnaires
* Patient with diabetic retinopathy

Min Age: 50 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge of AMD | throughout the study, 2 years at maximum
  Assesment concern patients knowledge of AMD disease, the treatment of AMD, the diagnostic of AMD and the knowledge on the AMD risk factors A 12 items standardised questionnaire will be used
Social vulnerability | throughout the study, 2 years at maximum
  Assessed by EPICES scale (Evaluation of Precariousness and Health Inequalities in the Health Examination Centers). It is an individual indicator of precariousness that takes into account the multidimensional nature of precariousness. Compsed of 11 items . 4 unfavorable answers indicate a Social vulnerability

SECONDARY OUTCOMES:
Health literacy. | throughout the study, 2 years at maximum
  Assessed by the Health Literacy Questionnaire (HLQ) scale. It has nine scales that each measure an aspect of the multidimensional construct of health literacy.
  Higher scores assess for an good health literacy

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Ophtalmologie, Limoges, France